CLINICAL TRIAL: NCT03971097
Title: The Effect of a Self-Forgiveness Model on Self-Stigma in Individuals Diagnosed With Substance Use Disorder.
Brief Title: The Effect of Self-Forgiveness on Self-Stigma in Addiction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Indiana University of Pennsylvania (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19030237
Record Dates: First submitted 2019-05-04; First posted 2019-06-03 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-01

CONDITIONS: Substance Use Disorders; Opiate Dependence; Opiate Withdrawal Syndrome; Opioid-use Disorder; Alcohol Withdrawal; Alcohol Abuse; Alcohol Use Disorder; Cocaine Abuse; Cocaine Use Disorder; Cocaine Withdrawal; Benzodiazepine Abuse; Benzodiazepine Dependence; Substance Abuse; Heroin Overdoses; Heroin Withdrawal; Heroin Abuse
Keywords: Substance abuse; Addiction; Opiates; Alcohol; Cocaine; Benzodiazepine; Heroin; Self-forgiveness; Self-stigma
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Alcoholism; Cocaine-Related Disorders; Heroin Dependence; Behavior, Addictive | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to examine differences between two groups of individuals receiving treatment at a residential drug and alcohol rehabilitation facility located at UPMC's McKeesport campus. The control group will receive treatment as usual (TAU) which includes group therapy, 12-step meetings facilitated by outside representatives of Alcoholics Anonymous (AA) and Narcotics Anonymous (NA), medical care, and individual needs assessment with recommendations for aftercare. The experimental group will receive TAU plus six additional individual counseling sessions that include integration of a self-forgiveness model developed by Worthington (2013). Differences between the groups will be measured by analyzing pre-test and post-test data on the Self-Forgiveness Dual Process Scale (SFDPS) (Griffin, Worthington, Davis, Hook, & Maguen, 2018) and the Substance Abuse Self-Stigma Scale (SASSS) (Luoma et al., 2013).
Who Masked: Participant
Masking Description: Participants will not be made aware of their status in either the control group or experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (TAU) (Active Comparator): Participants of the study who will receive the normal programming schedule or treatment as usual (TAU).
  Interventions: Behavioral: Treatment as Usual (TAU)
- Experimental Group (TAU plus self-forgiveness model) (Experimental): Participants of the study who will receive TAU plus six additional individual counseling sessions that include integration of a self-forgiveness model developed by Everett L. Worthington.
  Interventions: Behavioral: Six Step Model of Self-Forgiveness; Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Six Step Model of Self-Forgiveness — The six-step model includes a workbook that applies Worthington's (2013) conceptualization of self-forgiveness and guides the practitioner and participant through the self-forgiveness process. Each step provides a framework for techniques and includes psychoeducation, interventions, and "homework" to be completed in between sessions. The individual sessions will not conflict with the timing or content of the unit's regular treatment schedule, thus, participation in the study will not affect a patient's ability to participate in TAU. All interventions will be done individually to ensure that participant confidentiality is respected throughout the therapeutic process.
  Arms: Experimental Group (TAU plus self-forgiveness model)
Behavioral: Treatment as Usual (TAU) — Treatment as Usual (TAU) includes four group therapy sessions facilitated by the social services team (counselors and social workers), two 12-step meetings facilitated by outside representatives of Alcoholics Anonymous (AA) and Narcotics Anonymous (NA), dietary, spirituality, medical care including vital signs and the administration of prescribed medication by the nursing staff, and individual needs assessment with a recommendation of appropriate aftercare.

SUMMARY:
This study has an experimental design and will examine the difference in pre-test and post-test data on the Self-Forgiveness Dual Process Scale (SFDPS) (Griffin, Worthington, Davis, Hook, & Maguen, 2018) and the Substance Abuse Self-Stigma Scale (SASSS) (Luoma et al., 2013). Data will be collected from two groups of participants receiving counseling at the short-term rehabilitation facility located at University of Pittsburgh Medical Center's (UPMC). Individuals who agree to participate in the study will be randomly assigned to either the experimental group (EG) or the control group (CG). Data collected will include pre-test SFDPS and SASSS scores for the EG and the CG (collected within 24-hours of admission), and post-test SFDPS and SASSS scores for the EG and CG (collected after 14 days). ANCOVA will be used to analyze the pre-test and post-test data recorded from participants' scores.

DETAILED DESCRIPTION:
Participants of this study will consist of individuals 18 years of age or older, who have been admitted to the short-term rehabilitation program affiliated with UPMC and have agreed to take part in research designed to examine the relationship between self-forgiveness and self-stigma in individuals with SUD.

Patients will be made aware of the study by the principal investigator during an initial, in-person assessment that will occur within 48 hours of their admission to the unit. All patient rooms on this unit are limited to one patient which allows for privacy. Those who express interest, will be provided a copy of the Informed Consent Form and made aware of their right to decline participation or withdraw at any time, the limits of confidentiality, and that a lack of participation will not affect the level of care they receive. Patients who choose to participate in the study will be required to agree to the terms detailed in the consent form by signing and dating the form. Patients will then be assigned a participant number which be recorded on a link sheet only available to the principal investigator. Randomization software developed by GraphPad Software, Inc. will be used to randomly assign participants to either the experimental group or control group and that group assignment will be recorded on the link sheet. Participants will not be made aware of the group to which they have been assigned.

Prior to administering the SFPDS and SASSS to the participant, the principal investigator will write the corresponding participant number and group assignment on the top right-hand corner of the assessments. The participant will be asked to recall an event from their past that currently evokes feelings of regret. The participant will then be provided a copy of the SFDPS and SASSS. Because cultural and demographic factors such as level of education and physical disabilities are more common with this population, participants can choose to have the assessments administered orally. It is estimated that combined, the assessments will take 30 to 40 minutes to administer. To increase validity, participants will be informed that their answers will not be shared with other participants or members of the treatment team. Completed assessments will be collected and placed in an individual participant folder accessible only to the principal investigator. SFDPS and SASSS scores will be recorded on the link sheet in the pre-test columns.

Over the next 14 days, in addition to treatment as usual (TAU), participants in the experimental group will be introduced to techniques based on a six-step model of self-forgiveness during six individual sessions facilitated solely by the principal investigator. Participants in the control group will participate in the daily TAU schedule which includes four group therapy sessions facilitated by the social services team (counselors and social workers), two 12-step meetings facilitated by outside representatives of Alcoholics Anonymous (AA) and Narcotics Anonymous (NA), dietary, spirituality, medical care including vital signs and the administration of prescribed medication by the nursing staff, and individual needs assessment with a recommendation of appropriate aftercare. The six-step model includes a workbook that applies Worthington's conceptualization of self-forgiveness and guides the practitioner and participant through the self-forgiveness process. Each step provides a framework for techniques and includes psychoeducation, interventions, and "homework" to be completed in between sessions. The individual sessions will not conflict with the timing or content of the unit's regular treatment schedule, thus, participation in the study will not affect a patient's ability to participate in TAU. All interventions will be done individually to ensure that participant confidentiality is respected throughout the therapeutic process. After the sixth session, participants will be administered the SFDPS and SASSS for a second time. Scores will be recorded on the link sheet in the post-test columns. Participants who were in the control group will be offered a copy of the self-forgiveness workbook and provided additional support if requested.

Power analysis was performed utilizing G*Power 3.1, a stand-alone power analysis program for statistical tests used in the social, behavioral, and biomedical sciences. Using a desired power of .8 and a p-value of <.05, it was determined that an appropriate sample size to detect a significant difference in pre-test and post-test scores on the SFDPS and SASSS between the experimental group and control group is N=128 participants. Thus, the selection process will be repeated until a minimum of 64 experimental group participants and a minimum of 64 control group participants have completed the study.

The email sent to the social services team, the nursing staff, and the unit supervisors at UPMC McKeesport will ensure that the appropriate staff members at the facility are aware of the purpose of this study, the details of the Informed Consent, the content being assessed, and the nature of the workbook. Participants will be encouraged to follow up with the principal investigator or a staff member if they experience any distressing emotions related to their participation in the study. Having these staff members aware of the study and available to participants to process any issues that may arise from their participation will serve as a protective factor and mitigate potential risks. Participation in the study is strictly voluntary and each participant reserves the right to withdraw from the study at any time. Participation or non-participation in this study will not impact participant status in the program in any way. Participants will be notified of the limits of confidentiality and the mandated reporting role of the principal investigator during the Informed Consent process. As the participants will be provided with a copy of the Informed Consent Form, they will be able to refer to this information on their own at any time.

The initial assessments, informed consent process, and workbook sessions will be conducted either in a private hospital room or a confidential group room setting to protect the privacy of study participants. The principal investigator's notes, scores from the SFDPS and SASSS, and answers from the workbook exercises (together referred to as "data") will be confidential and none of the information gathered during these meetings will be discussed or shared with staff members at the facility. Once the informed consent process is complete, participants will be assigned a number that will correspond to their data. The principal investigator will create a "link sheet" that will connect the participant's name (provided on the consent form) with the number on the notes, scoring sheets, and workbook. This sheet will only be seen by the principal investigator and will be destroyed upon completion of the study. As participants complete the study, their names will be removed from the link sheet. Prior to analysis of the data, no one apart from the principal investigator will have access to the data. All information gathered, analyzed, and reported will be presented in aggregate form so that no identifying characteristics can be made. Any data that is collected will be also be secured electronically via password and encryption or physically in a locked filing cabinet in a secured office.

There are no guaranteed benefits for participating in this study; however, participants may experience a reduction in the guilt, shame, and self-blame that often accompanies addiction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Admitted to the short-term rehabilitation program at UPMC McKeesport.
* Have agreed to take part in research designed to examine the relationship between self-forgiveness and self-stigma in individuals with SUD.

Exclusion Criteria:

• Patients who previously took part in the study, were discharged, and then readmitted to the unit within six months due to relapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Substance Abuse Self-Stigma Scale (SASSS) | 14 days
  Self-stigma can be defined as internalized stigma and is closely related to shame. The SASSS is a 40-item assessment (minimum total score is 40; maximum total score is 200) based on relational frame theory and is designed to measure self-stigma experienced by individuals who are misusing substances. It contains four discrete subscales and asks the participant to indicate on a 5-point Likert scale the frequency of thoughts/experiences, how much people would react to them, and the degree to which a true statement characterizes them. Higher scores reflect higher levels of self-stigma. The four subscales include self-devaluation (8 items; min score 8; max score 40), fear of enacted stigma (9 items; min score 9; max score 45), stigma avoidance (13 items; min score 13; max score 65), and values disengagement (10 items; min score 10; max score 50).
Self-Forgiveness Dual Process Scale (SFDPS) | 14 days
  The SFDPS is a 10-item assessment (minimum total score is 10; maximum score is 70) based on social cognitive theory and contains two subscales, values reorientation and esteem restoration. Responses are measured on a 7-point Likert scale ranging from strongly disagree to strongly agree. Higher scores reflect higher levels of self-forgiveness. The first five questions (5 items; min score 5; max score 35) focus on reorientation toward positive values and measure the cognitive shift toward accepting responsibility for one's perceived offense and committing to align future behavior with positive values. The second five questions (5 items; min score 7, max score 35) focus on restoring one's person sense of self-esteem and measure the extent to which one has replaced self-condemning emotions with self-affirming ones.

CONTACTS AND LOCATIONS:
Overall Officials: Holly P Branthoover, EdD., Study Chair — Indiana University of Pennsylvania; Michael P Verona, MA, Principal Investigator — Indiana University of Pennsylvania
Locations (1):
- UPMC McKeesport, McKeesport, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
All information gathered, analyzed, and reported will be presented in aggregate form and exclude identifying characteristics.

REFERENCES:
- [Background] Griffin BJ, Worthington EL, Davis DE, Hook JN, Maguen S. Development of the Self-Forgiveness Dual-Process Scale. J Couns Psychol. 2018 Nov;65(6):715-726. doi: 10.1037/cou0000293. PMID 30421952
- [Background] Luoma JB, Nobles RH, Drake CE, Hayes SC, O'Hair A, Fletcher L, Kohlenberg BS. Self-Stigma in Substance Abuse: Development of a New Measure. J Psychopathol Behav Assess. 2013 Jun 1;35(2):223-234. doi: 10.1007/s10862-012-9323-4. PMID 23772099
- [Background] Worthington, E.L. (2013) Moving forward: Six steps to forgiving yourself and breaking free from the past. New York, NY: Waterbrook.